CLINICAL TRIAL: NCT05319119
Title: The Impact Of Revascularization Related By Blood Fractional Flow Reserve Calculated By Coronary Artery CTA On Prognosis
Brief Title: Fractional Flow Reserve Derived From CT Related Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Chuanyu Gao, Professor, Henan Institute of Cardiovascular Epidemiology
Other Study IDs: BHe
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Coronary Angiography; Fractional Flow Reserve, Myocardial; Coronary Artery Disease
Keywords: Fractional Flow Reserve; CT-FFR; prognosis; coronary Revascularization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1.CT-FFR Related Group: Coronary diseased artery CTFFR>80%, secondary prevention of coronary heart disease;Coronary diseased artery CTFFR≤80% revascularization at the lesion site and regular medication after PCI
- Coronary Angiography Related Group: Coronary diseased artery CTFFR≤80%, coronary angiography decision does not require revascularization but apply coronary heart disease secondary prevention medication;Coronary diseased artery CTFFR>80%,However, revascularization was performed according to conventional angiographic decisions and postoperative regular service was performed.For multivessel disease, although coronary revascularization is performed, there are still diseased artery with CTFFR≤80% and no revascularization is performed.

SUMMARY:
This study is a retrospective, single-center study.This experiment aims to explore the influence of CT-FFR as a relevant for revascularization on the prognosis of patients with coronary heart disease, assessing concurrent on different basis the difference of prognosis of patients with revascularization was analyzed, and the significance of revascularization related by CT-FFR was analyzed.This study is a retrospective study. The treatment strategies of all patients are based on the results of CAG，including coronary revascularization.After calculating the CT-FFR value, the above doctors will formulate treatment strategies based on the results and formulate treatment strategies retrospectively.

DETAILED DESCRIPTION:
Research Objects and Criteria:Patients who had undergone coronary angiography and Coronary Artery CTA in Fuwai Central China Cardiovascular Hospital.Preliminary screening of patients is carried out in the medical record system, CT imaging workstation, and interventional center imaging workstation to confirm data integrity.

Standard constrain:①Diagnosed or suspected coronary heart disease patients during the diagnosis and treatment process.②From December 2017 to December 2020, coronary artery CTA and coronary angiography were performed simultaneously in Fuwai Central China Cardiovascular Hospital. (coronary artery CTA before the coronary angiography, but no more than 28 days apart).③Age 18 to 75 years old.

Exclusion criteria:①Severe artefacts, misalignment, or calcifications in coronary CTA images affect CT-FFR measurements.② Contraindications to antiplatelet drugs③ Patients with acute myocardial infarction within 6 months.④ PCI or CABG or heart transplantation and other operations that may affect the outcome⑤ Severe heart failure⑥ Pregnant patients⑦ Combined tumor patients⑧ Have a history of other serious heart disease⑨Contraindications to coronary angiography drop out standard:① Abnormal research results ② Failure to achieve the expected therapeutic effect due to other serious diseases ③ Violation of the research plan④ Lost to follow-up ⑤ The relevant data is seriously missing, which affects the experimental data

Case grouping method:

1. CT-FFR related Group:①Coronary diseased artery CTFFR>80%, secondary prevention of coronary heart disease ② Coronary diseased artery CTFFR≤80% revascularization at the lesion site and regular medication after PCI
2. Coronary angiography related Group:①Coronary diseased artery CTFFR≤80%, coronary angiography decision does not require revascularization but apply coronary heart disease secondary prevention medication. ②Coronary diseased artery CTFFR>80%,However, revascularization was performed according to conventional angiographic decisions and postoperative regular service was performed.For multivessel disease, although coronary revascularization is performed, there are still diseased artery with CTFFR≤80% and no revascularization is performed.

End point：①Primary endpoint: all-cause death/cardiac death,②Secondary endpoints:myocardial infarction, target vessel repeat revascularization, brain stroke readmission for cardiovascular events, abnormal laboratory tests, new-onset heart failure, or progression to severe heart failure Statistics and analysis of research data：The data collected in the group at different recording times are selected if they satisfy the normal distribution.

Repeated measures ANOVA; if normal distribution is not met, rank sum test is used.The data between groups were analyzed by one-way analysis of variance. For count data (include rate) use X² or Fisher's exact probability test.Statistically significant at p < 0.05 Use the Kaplan-Meier method to describe the survival rate of each group and draw the survival curve, and then use the Log-rank Test Calculate the test statistic, with p < 0.05 as statistically significant.The factor p < 0.05 obtained from the univariate Cox analysis was included in the multivariate Cox proportional wind in the risk model, hazard ratios, 95% confidence intervals were calculated and multivariate adjustment analysis was performed. Take p < 0.05 as having statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* ①Diagnosed or suspected coronary heart disease patients during the diagnosis and treatment process

  * From December 2017 to December 2020, coronary CTA and coronary artery CTA were performed simultaneously in Huazhong Fuwai Hospital.

Patients with CAG (coronary CTA before coronary angiography after CAG, no more than 28 days apart).

③Age 18 to 75 years old.

Exclusion Criteria:

* ① The presence of severe artifact, dislocation or calcification in coronary CTA images affects FFRCT measurement. ② Contraindications to antiplatelet drugs

  * Patients with acute myocardial infarction within 6 months④ PCI or CABG or heart transplantation and other operations that may affect the outcome ⑤ Severe heart failure⑥ Pregnant patients⑦ Combined tumor patients⑧ Life expectancy < 2 years⑨ Have a history of other serious heart disease⑩ Contraindications for CAG⑪ Not suitable to participate in this researcher due to other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed or suspected coronary heart disease patients with typical symptoms or objective evidence of ischemia such as ECG, exercise treadmill, coronary CTA or CAG
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-04-06 (Estimated); Study Completion 2022-04-29 (Estimated)

PRIMARY OUTCOMES:
All-cause death or Myocardial infarction | 1 year
  Cardiovascular, non-cardiovascular and undetermined death or Target vessel related and non-target vessel related MI

SECONDARY OUTCOMES:
Heart failure | 1 year,2 years
  Heart failure
Non-target vessel revascularization | 1 year,2 years
  The ischemia driven and non-ischemia driven non-target vessel revascularization
Cardiac death | 1 year,2 years
  Cardiovascular death
Target vessel revascularization | 1 year,2 years
  The ischemia driven and non-ischemia driven target vessel revascularization
Myocardial infarction | 1 year,2 years
  Target vessel related and non-target vessel related MI
Stroke | 1 year,2 years
  Stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China